CLINICAL TRIAL: NCT05741710
Title: A Pilot Study to Assess the Use of Methylone in the Treatment of PTSD IMPACT-1 (Investigation of Methylone for Post-Traumatic Stress Disorder [PTSD])
Brief Title: A Study to Assess the Use of Methylone in the Treatment of PTSD
Acronym: IMPACT-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Transcend Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TT-TSND-201
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Post Traumatic Stress Disorder
Keywords: methylone; PTSD; IMPACT-1; Transcend Therapeutics
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — methylone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylone (Experimental)
  Interventions: Drug: Methylone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylone — Methylone capsules, given orally, once a week for 4 weeks
  Arms: Methylone
Drug: Placebo — Placebo capsules to match methylone, given orally, once a week for 4 weeks. NOTE: Placebo is only in Part B
  Arms: Placebo

SUMMARY:
This study is evaluating the safety, tolerability, and efficacy of methylone in adults with PTSD. The study will be conducted in two parts.

* Part A is open-label and will enroll up to 15 participants with PTSD
* Part B is randomized (1:1), double-blind, placebo-controlled and will enroll up to 64 participants with PTSD

Eligible participants will enter a 4-week Treatment Period where they will receive methylone once weekly for 4 weeks (4 treatment sessions). Following the Treatment Period, participants will enter a 6-week Follow-up Period which includes 3 reflection visits (Week 4, 5, and 6) and a final study visit at Week 10.

ELIGIBILITY:
Inclusion Criteria:

* Meets the DSM-5 criteria for current moderate to severe PTSD diagnosis, with a symptom duration of at least 6 months
* CAPS-5 score of ≥35 at Screening.
* Failed at least one treatment for PTSD (either psychotherapy or pharmacological treatment).
* Proficient in reading and writing in local language sufficient to complete questionnaires.
* Free from any other clinically significant illness or disease

Exclusion Criteria:

* Primary diagnosis of any other DSM-5 disorder
* Body mass index (BMI) <18 kg/m2 or ≥40 kg/m2.
* Smokes an average of >10 cigarettes and/or e-cigarettes per day
* Uncontrolled hypertension at Screening
* Use of a psychedelic (e.g., LSD, psilocybin, DMT, mescaline), or entactogens such as MDMA, within 12 months of Screening.
* Use of an SSRI or other antidepressant within 8 weeks of screening.
* Current or previous history of clinically significant cardiovascular/cerebrovascular conditions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Clinician-Administered PTSD Scale for the DSM-5 (CAPS-5) total severity score | up to 10 weeks
  CAPS-5 is a structured interview designed to assess PTSD symptoms severity. The total severity score ranges from 0 to 80, with a higher score indicating more severe symptoms.

SECONDARY OUTCOMES:
Change from Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) total score | up to 10 weeks
  The MADRS is a 10-item, clinician-rated scale designed to assess severity of depression. The total score ranges from 0 to 60, with a higher score indicating more severe depression.
Change from Baseline in PTSD Checklist for DSM-5 (PCL-5) | up to 10 weeks
  The PCL-5 is a 20-item, patient-rated scale designed to measure severity of PTSD symptoms. The total score ranges from 0 to 80, with a higher score indicating more severe PTSD symptoms.
Change from Baseline in Sheehan Disability Scale (SDS) | up to 10 weeks
  The SDS is a 3-item, patient-rated scale designed to measure disability and impairment across three domains: work/school, social life, and family life / home responsibilities. Each domain is scored from 0 to 10, with higher scores represented more disability. Total sores range from 0 to 30.
Incidence of treatment-emergent adverse events (TEAEs) | up to 10 weeks
  Type and rates of adverse events

CONTACTS AND LOCATIONS:
Locations (16):
- United States (8):
  - Mountain View Clinical Research, Denver, Colorado
  - Clinical Neuroscience Solutions - Jacksonville, Jacksonville, Florida
  - Accel Research Sites, Maitland, Florida
  - Sunstone Therapies, Rockville, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Cenexel HRI, Berlin, New Jersey
  - The Rivus Wellness & Research Institute, Oklahoma City, Oklahoma
  - Cedar Clinical Research, Murray, Utah
- Ireland (2):
  - Tallaght Adult Mental Health Services, Dublin
  - La Nua Day Hospital Mental Health Centre, Galway
- United Kingdom (6):
  - Mirabilis Health, Belfast, Northern Ireland
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Glasgow Clinical Research Facility, QEUH, Glasgow
  - Clerkenwell Health, London
  - King's College, London
  - Oxford Health NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No